CLINICAL TRIAL: NCT04871347
Title: A Multi-center, Phase Ia/Ib, Open Clinical Study to Evaluate the Safety and Efficacy of TWP-101 in Patients With Advanced Solid Tumor
Brief Title: The Safety and Efficacy of TWP-101 in Patients With Advanced Solid Tumor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong TheraWisdom Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TWP-101-12
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-05

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Cohort (Experimental): Three dose levels of TWP-101 will be tested by a conventional 3 + 3 study design.
  Interventions: Drug: TWP-101
- Dose Expansion Cohort (Experimental): Once the effective dose has been determined, an expansion cohort will be opened to evaluate the efficacy and safety of the selected dose.
  Interventions: Drug: TWP-101

INTERVENTIONS:
Drug: TWP-101 — IV infusion
  Other Names: Sytalizumab Injection

SUMMARY:
This is a multi-center, phase Ia/Ib, open clinical study to evaluate the safety and efficacy of TWP-101 in patients with advanced solid tumor. This study consists of two parts (Part A and Part B). Part A was a dose escalation study, and Part B was a dose expansion study.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically or cytologically confirmed advanced solid tumor that failed, couldn't tolerate or refused standard treatments;
* ECOG score 0 or 1;
* At least 1 measurable lesion according to RECIST 1.1

Exclusion Criteria:

* Known hypersensitivity to any ingredient of TWP-101;
* Receiving any anti-cancer drugs within 4 weeks;
* History of serious systemic diseases;
* History of serious autoimmune diseases;
* Pregnancy or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2021-08-30 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) | From the first dose of study drug up to 4 weeks
Incidence of adverse events and serious adverse event (defined by the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE V5.0)) and irAE. | From enrollment until 90 days after the last dose

SECONDARY OUTCOMES:
Objective Response Rate (ORR) by RECIST Version 1.1 | From first dose to disease progression or end of study, an average of 2 years
Duration of Response (DOR) | From first dose to disease progression, an average of 2 years
Disease control rate (DCR). | From first dose to disease progression or end of study, an average of 2 years
Progression free survival (PFS). | From first dose to disease progression or end of study, an average of 2 years
Maximum measured plasma concentration (Cmax) of TWP-101. | From first dose until 90 days after the last dose
Time to maximum plasma concentration (Tmax) of TWP-101. | From first dose until 90 days after the last dose
Half-life (T1/2) of TWP-101. | From first dose until 90 days after the last dose
Immunogenicity profile of TWP-101. | From first dose until 90 days after the last dose
  Blood samples will be collected from subjects post treatment for assessment to detect the presence of anti-drug antibodies and neutralizing antibodies by meso scale discovery(MSD).

CONTACTS AND LOCATIONS:
Locations (1):
- Harbin Medical University Cancer Hospital, Harbin, Heilongjiang, China